CLINICAL TRIAL: NCT02009605
Title: An Open-label, Single-armed Pilot Study to Evaluate the Efficacy of Icotinib in Previously Treated Non/Light-smoking Patients With Squamous Lung Cancer
Brief Title: Icotinib in Previously Treated Non/Light-smoking Patients With Advanced Squamous Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Qiong Zhao, Prof., Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYTOP 1401
Record Dates: First submitted 2013-12-08; First posted 2013-12-12 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Squamous Cell Carcinoma of Lung
Keywords: icotinib, SCC
MeSH Terms: interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- one arm (Experimental): Icotinib of routine dose Icotinib: 125mg, oral administration, three times per day.
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — 125mg, oral administration, three times per day.
  Other Names: BPI-2009

SUMMARY:
This study is designed to evaluate the efficacy of icotinib at routine dose in previously treated non/light-smoking patients with advanced squamous cell lung cancer.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy of icotinib at routine dose in previously treated non/light-smoking patients with advanced squamous cell lung cancer. An objective response (OR) was defined as a patient having a best overall response of either complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors, confirmed at least 28 days following the date of the initial response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic or recurrent squamous cell lung cancer from the primary lesion and/or lymph nodes, stage IIIB or IV patients with non-smoking or light-smoking history.
* Failure of at least 1, and no more than 2, prior chemotherapy regimens for advanced disease (either due to progressive disease or toxicity).
* Have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan.
* Be >= 18 years of age.
* Expected survival period over 12 weeks;
* ECOG PS 0-2. Adequate organ system function as defined within the protocol.
* Patients with a history of CNS metastases or cord compression are allowed if they have been definitively treated and are clinically stable.
* Consent compliance research plan and follow-up process, and be able to carry out oral therapy; Provision of written informed consent.
* In women of childbearing age, must be in before starting treatment within 7 day of urine pregnancy test and the result is negative, and not in the lactation period, and reproductive age men and women prior to entry into the study, the research process until 90 days after stopping all agree to use reliable methods of contraception;
* Weight loss =< 10% in past 6 months.
* Adequate tumor tissue for detection of molecular biomarkers.

Exclusion Criteria:

* Patients who have previously received treatment with EGFR-TKIs.
* Concomitant treatment with any other experimental drug under investigation or anti-tumor therapy;
* Symptomatic CNS metastases or newly diagnosed CNS metastases that have not yet been definitively treated with radiation and/or surgery.
* Known severe hypersensitivity to icotinib or any of the excipients of this product.
* Presence of uncontrolled pleural effusion or/and peritoneal effusion;
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study.
* Past or current history of neoplasm (other than the entry diagnosis) in past 5 years, with the exception of treated basal cell carcinoma or carcinoma in situ of the cervix, or other cancers cured by local therapy alone.
* Women who are lactating.or have positive pregnancy test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 4 Weeks
  Number of participants with an objective response. An objective response (OR) was defined as a patient having a best overall response of either complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors, confirmed at least 28 days following the date of the initial response.

SECONDARY OUTCOMES:
Progression free survival | 3 months
  Progression free survival was defined as the time from the date of first dose of study medication to the date of first documentation of tumor progression or death due to any cause, whichever occurred first.
Overall survival | 14 months
  Overall Survival was assessed via calculation of the time to death due to any cause. If a participant was known to have died, the time to death was defined as the time from the date of randomization to the date of death. Otherwise, a participant was censored at the last date they were known to be alive.
Number of Participants with Adverse Events | 3 months
  Adverse events, serious adverse events, incidence of and reason for study drug dose interruptions and discontinuations, laboratory assessments, vital signs.

OTHER OUTCOMES:
Life quality | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Qiong, Dr., Principal Investigator — Zhejiang University
Locations (1):
- 79 Qingchun Road, Hangzhou, Zhejiang, China